CLINICAL TRIAL: NCT04424251
Title: A Randomized, Double-blind, Placebo-controlled, Two-stage Phase II Study Evaluating the Efficacy and Safety of HSK21542 in Inducing Postoperative Analgesia in Subjects Undergoing Elective Laparoscopic Surgery Under General Anesthesia
Brief Title: Efficacy and Safety of HSK21542 in Inducing Postoperative Analgesia in Undergoing Elective Laparoscopic Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK21542-201
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- stage I：HSK21542 0.4 μg/kg (Experimental): Preoperative:0.4 μg/kg Postoperative:0.2 μg/kg； intravenous injection
  Interventions: Drug: Experimental: stage I：HSK21542 0.4 μg/kg
- stage I：HSK21542 1 μg/kg (Experimental): Preoperative:1 μg/kg Postoperative:0.5 μg/kg；intravenous injection
  Interventions: Drug: Experimental: stage I：HSK21542 1 μg/kg
- stage I：HSK21542 0.5μg/kg (Experimental): Postoperative: 0.5μg/kg；intravenous injection
  Interventions: Drug: Experimental: stage I：HSK21542 0.5μg/kg
- stage I：HSK21542 1μg/kg (Experimental): Postoperative: 1μg/kg；intravenous injection
  Interventions: Drug: Experimental: stage I：HSK21542 1μg/kg
- stage II：HSK21542 0.5μg/kg (Experimental): Postoperative: 0.5μg/kg；intravenous injection
  Interventions: Drug: Experimental: stage II：HSK21542 0.5μg/kg
- stage II：HSK21542 1μg/kg (Experimental): Postoperative: 1μg/kg；intravenous injection
  Interventions: Drug: Experimental: stage II：HSK21542 1μg/kg
- Postoperative: Placebo (Placebo Comparator): Placebo；intravenous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Experimental: stage I：HSK21542 0.4 μg/kg — Once preoperative and once each at 0, 8, and 16 h postoperative, for a total of 4 administrations
  Arms: stage I：HSK21542 0.4 μg/kg
Drug: Experimental: stage I：HSK21542 1 μg/kg — Once preoperative and once each at 0, 8, and 16 h postoperative, for a total of 4 administrations
  Arms: stage I：HSK21542 1 μg/kg
Drug: Experimental: stage I：HSK21542 0.5μg/kg — once each at 0, 8, and 16 h postoperative, for a total of 3 administrations
  Arms: stage I：HSK21542 0.5μg/kg
Drug: Experimental: stage I：HSK21542 1μg/kg — once each at 0, 8, and 16 h postoperative, for a total of 3 administrations
  Arms: stage I：HSK21542 1μg/kg
Drug: Experimental: stage II：HSK21542 0.5μg/kg — once each at 0, 8, and 16 h postoperative, for a total of 3 administrations
  Arms: stage II：HSK21542 0.5μg/kg
Drug: Experimental: stage II：HSK21542 1μg/kg — once each at 0, 8, and 16 h postoperative, for a total of 3 administrations
  Arms: stage II：HSK21542 1μg/kg
Drug: Placebo — once each at 0, 8, and 16 h postoperative, for a total of 3 administrations
  Arms: Postoperative: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, two-stage phase II clinical study. The main objective is to evaluate the efficacy and safety of HSK21542 injection and explore the recommended dose and administration frequency for subsequent Phase II studies in conjunction with the pharmacodynamic (PD) and pharmacokinetic (PK) characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. 18 ≤ age ≤ 70 years old, with no gender requirement
2. American Society of Anesthesiologists (ASA) Class I-II
3. 18 kg/m^2 ≤ BMI ≤ 40 kg/m^2
4. Subjects undergoing elective laparoscopic surgery under general anesthesia with an expected surgery duration of 1-5 h (inclusive)
5. Agree to participate in this trial and voluntarily sign the informed consent form;

Exclusion Criteria:

1. History of allergy to opioids, such as urticaria, or allergic to the intraoperative anesthetics prescribed in the protocol;
2. History or evidence of any one of the following diseases prior to screening:

   1. History of cardiovascular diseases: Uncontrolled hypertension (systolic blood pressure [SBP] ≥ 170 mmHg and/or diastolic blood pressure [DBP] ≥ 105 without antihypertensive treatment, or SBP > 160 mmHg and/or DBP > 100 mmHg despite antihypertensive treatment), aneurysm, severe arrhythmia, heart failure, Adams-Stokes syndrome, New York Heart Association (NYHA) Class ≥ III, severe superior vena caval syndrome, pericardial effusion, acute myocardial ischemia, unstable angina, myocardial infarction in the last 6 months before screening, history of tachycardia/bradycardia requiring medication, and II-III degree atrioventricular block (excluding patients with pacemakers);
   2. History of respiratory disorder: Severe chronic obstructive pulmonary disease, acute exacerbation of chronic obstructive pulmonary disease, severe bronchostenosis, throat mass, history of (bronchial) tracheoesophageal fistula or airway tear, and severe respiratory tract infection in the last 2 weeks before screening;
   3. History of disorders in the nervous and psychiatric system: History of craniocerebral injury, possible convulsions, intracranial hypertension, cerebral aneurysms, and history of cerebrovascular accidents; history of schizophrenia, mania, mental aberration, long-term use of psychotropic drugs, and cognitive disorder; history of depression, anxiety, and epilepsy, etc.;
   4. Underwent major surgery within 3 months before screening and was judged by the investigator to have potential effect on the postoperative pain evaluation;
3. Any of the following airway management risks during screening:

   1. Acute asthma attacks;
   2. Sleep apnea syndrome;
   3. History or family history of malignant hyperthermia;
   4. History of failed tracheal intubation;
   5. Difficult airway (modified Mallampati score ≥ III) as determined by the investigator;
4. In receipt of any of the following drugs or therapies during the screening period:

   1. The time between randomization and the last dose of opioid or non-opioid (such as acetaminophen, aspirin [daily dose of > 100 mg], indomethacin, diclofenac, parecoxib sodium and other non-steroidal anti-inflammatory drugs) analgesics is shorter than 5 half-lives of the drug or the duration of drug efficacy (whichever is longer);
   2. Continuous use of opioid analgesics for more than 10 days for any reason within 3 months before screening;
   3. Use of drugs that affect the analgesic effect within 14 days before randomization, including but not limited to: Sedative hypnotics (benzodiazepines [triazolam, diazepam, midazolam, etc.], non-benzodiazepines [zolpidem, zopiclone, zaleplon, etc.]), sedative anesthetics (sevoflurane, anesthesia ether, nitrous oxide, thiopental, ketamine, etomidate, etc.), glucocorticoids (dexamethasone hydrochloride , methylprednisolone, etc.), anti-epilepsy drugs (carbamazepine, sodium valproate, etc.), anxiolytics (carbamazepine, diazepam, etc.), antidepressants (imipramine, amitriptyline, etc.), and Chinese herbal medicines or Chinese patent medicines with analgesic and sedative effects;
   4. Expected to receive anti-tumor drugs and treatments during the period from 14 days before randomization to the end of the follow-up period, including but not limited to chemotherapeutic drugs, targeted drugs, and Chinese herbal medicines.
   5. The time between randomization and the last use of diuretics and compound drugs containing diuretic components is shorter than 5 half-lives of the drug or the duration of drug efficacy (whichever is longer);
5. Laboratory test parameters meet one of the following criteria in the screening period and is confirmed by retests:

   1. White blood cell count < 3.0 x 10^9/L;
   2. Platelet count < 80 x 10^9/L;
   3. Hemoglobin <70 g/L;
   4. Prothrombin time > 1.5 x ULN;
   5. Activated partial thromboplastin time > 1.5 x ULN;
   6. Alanine aminotransferase and/or aspartate aminotransferase > 2 x ULN;
   7. Total bilirubin > 1.5 x ULN;
   8. Blood creatinine > 1.5 x ULN;
   9. Fasting blood glucose ≥ 11.1 mmol/L;
6. Without oxygen supplement during the screening period, the pulse oxygen saturation is < 92%;
7. During the screening period, the virological examination for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), treponema pallidum antibody, or human immunodeficiency virus (HIV) antibody is positive;
8. History of drug abuse, narcotics use and/or alcohol abuse within 3 months before screening. Alcohol abuse is defined as > 2 units of alcohol consumption per day (1 unit = 360 mL of beer containing 5% alcohol, 45 mL of liquor containing 40% alcohol, or 150 mL of wine);
9. Donated or lost ≥ 400 mL of blood within 3 months before screening;
10. Participated in any drug clinical trials within 3 months before screening (defined as the administration of the investigational product or placebo);
11. Women who are pregnant or breastfeeding; fertile women or men who are unwilling to use contraception during the trial; subjects who are planning pregnancy within 3 month after the completion of the trial (including male subjects);
12. Subjects determined by the investigator to be unsuitable for participating in this clinical study for any other reason.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Sum of Pain Intensity Differences (SPID) | Frome administration until 24 hours after administration
  The time-weighted SPID at rest within 0-24 h after the first postoperative administration in each group

SECONDARY OUTCOMES:
Sum of Pain Intensity Differences (SPID) | Frome administration until 24 hours after administration
  The time-weighted sum of pain intensity differences of the rest pain in each group within 0-12 h after the first postoperative dose
Use of remedial analgesics | Frome administration until 24 hours after administration
  Cumulative dose of remedial analgesics (mg of morphine injection) in each group within 0-12 h and 0-24 h after the first postoperative dose, the percentage of subjects in each group who have not used remedial analgesics, and the time to start using remedial analgesics
Pain Intensity Differences（PID） | Frome administration until 24 hours after administration
  The PID at rest at each scoring time point after the first postoperative administration in each group
The proportion of subjects with a NRS of ≤ 3 | Frome administration until 24 hours after administration
  The proportion of subjects in each group with a resting pain NRS of ≤ 3 at 12 h and 24 h after the first postoperative dose
Duration of analgesia | Frome administration until 24 hours after administration
  The duration of analgesia after the first postoperative administration in each group
Satisfaction scores on postoperative analgesia | Frome administration until 24 hours after administration
  Subject satisfaction score and investigator satisfaction score on postoperative analgesia at 24 h after the first postoperative administration in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, China

REFERENCES:
- [Derived] Zhong Y, Wang H, Yan M, Yang M, Zhang J, Nan L, Wang Z, Yang J, Wu J, Guo Q, Hu X, Xu H, Xu Q, Wang D. Efficacy and safety of peripherally-restricted kappa-opioid receptor agonist-HSK21542 for postoperative analgesia in patients undergoing laparoscopic abdominal surgery: a randomized, placebo-controlled phase 2 trial. Front Med (Lausanne). 2025 Jul 24;12:1604790. doi: 10.3389/fmed.2025.1604790. eCollection 2025. PMID 40776930